CLINICAL TRIAL: NCT00189917
Title: An Open-label, Controlled Phase I Pilot Study to Evaluate Safety and Immunogenicity of MVA-BN® Smallpox Vaccine in 18-40 Year Old Vaccinia-naïve Subjects With Atopic Disorders
Brief Title: Safety, Tolerability and Immune Response of IMVAMUNE (MVA-BN)Smallpox Vaccine in Patients With Atopic Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: POX-MVA-007; N01-AI-30016 (Other Grant/Funding Number: NIAID)
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Dermatitis, Atopic; Hay Fever
MeSH Terms: conditions — Dermatitis, Atopic; Rhinitis, Allergic, Seasonal | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

ARMS (4):
- GP 1: healthy, no AD (Experimental): Healthy subjects without any history of, or current signs and symptoms of atopic disease, receiving two doses IMVAMUNE (MVA-BN), subcutaneous.
  Interventions: Biological: IMVAMUNE (MVA-BN)
- GP2: prev. allerg. rhinitis (Experimental): Subjects having documentation of at least one allergic rhinitis event during the previous year, receiving two doses IMVAMUNE (MVA-BN), subcutaneous..
  Interventions: Biological: IMVAMUNE (MVA-BN)
- GP3: history of AD (Experimental): Subjects having documentation of a history of Atopic Dermatitis, receiving two doses IMVAMUNE (MVA-BN), subcutaneous..
  Interventions: Biological: IMVAMUNE (MVA-BN)
- GP4: active AD (Experimental): Subjects presenting active Atopic Dermatitis and having an individual SCORAD value between 1 and 15, receiving two doses IMVAMUNE (MVA-BN), subcutaneous.
  Interventions: Biological: IMVAMUNE (MVA-BN)

INTERVENTIONS:
Biological: IMVAMUNE (MVA-BN) — 1x10E08 TCID50, subcutaneous vaccination

SUMMARY:
The purpose of this study is to gather information on the safety and immunogenicity of an investigational smallpox vaccine in populations with atopic disorders.

ELIGIBILITY:
Inclusion Criteria:

All subjects

* Age 18-40.
* Read, signed and dated informed consent.
* Women of childbearing potential must use an acceptable method of contraception

Group 1: Healthy subjects

* No history of atopic dermatitis as documented in the patient file
* No active atopic dermatitis
* No other atopic disorders such as asthma or allergic rhinitis.
* Prick test without clinical significance
* IgE within normal range

Group 2: Subjects with history of atopic dermatitis

Group 3: Subjects with mild active atopic dermatitis

- SCORAD 1 - 15.

Group 4: Subjects with mild allergic rhinitis

* At least one active allergic rhinitis phase during last year.

Exclusion Criteria:

* Known or suspected history of smallpox vaccination or typical vaccinia scar.
* Positive test result in MVA specific ELISA at screening.
* Positive result in HIV or HCV antibody test at screening.
* Surface antigen of Hepatitis B Virus (HBsAg) positive at screening.
* Pregnant or breast-feeding women.
* Positive pregnancy test at screening and/or within 24 hours prior to vaccination.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) above the institutional upper limit of normal.
* Positive urine glucose by dipstick or urine analysis.
* Inadequate renal function defined as a serum creatinine above the institutional upper limit of normal; urine protein >30 mg/dl or trace proteinuria (by urine analysis or dipstick); and a calculated creatinine clearance <80 ml/min.
* Electrocardiogram (ECG) with clinical significance.
* Hemoglobin <11 g/dl; White blood cells less than 2,500 and more than 11,000/mm3; Platelets less than 140,000/mm3.
* Uncontrolled serious infection i.e. not responding to antimicrobial therapy.
* History of any serious medical condition, which in the opinion of the investigator would compromise the safety of the subject.
* History of or active autoimmune disease.
* Known or suspected impairment of immunologic function including, but not limited to, clinically significant liver disease; diabetes mellitus; moderate to severe kidney impairment.
* History of malignancy.
* History or clinical manifestation of clinically significant mental illness or haematological, renal, hepatic, pulmonary, central nervous, cardiovascular or gastrointestinal disorders.
* Any condition which might interfere with study objectives.
* History of immunodeficiency.
* History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, or other heart condition under the care of a doctor.
* Three or more of the following risk factors: High blood pressure, high blood cholesterol, diabetes mellitus or high blood sugar, a first degree relative who had a heart condition before the age of 50, smoking cigarettes.
* History of chronic alcohol abuse and/or intravenous drug abuse.
* History of allergic reactions likely to be exacerbated by any component of the vaccine.
* History of anaphylaxis or severe allergic reaction.
* Acute disease (illness with or without a fever) at the time of enrollment.
* Any vaccinations within a period starting 30 days prior to administration of the vaccine and ending at study conclusion.
* Chronic administration of immuno-suppressant or immune-modifying drugs.
* Post organ transplant subjects whether or not receiving chronic immunosuppressive therapy.
* Administration or planned administration of immunoglobulins and/or any blood -- Use of any investigational or non-registered drug.
* Blood donation 8 weeks in advance or during study participation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2004-04 (Actual); Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Occurrence, relationship and intensity of any serious adverse event at any time during the study.

SECONDARY OUTCOMES:
ELISA specific seroconversion rates and geometric mean titres (at all blood sampling time points).
Neutralisation assay specific seroconversion rates and geometric mean titres (at all blood sampling time points).

CONTACTS AND LOCATIONS:
Overall Officials: Frank von Sonnenburg, M.D., Principal Investigator — Department of Infectious Diseases and Tropical Medicine of the University of Munich
Locations (1):
- Department of Infectious Diseases and Tropical Medicine, Munich, Bavaria, Germany

REFERENCES:
- [Result] von Sonnenburg F, Perona P, Darsow U, Ring J, von Krempelhuber A, Vollmar J, Roesch S, Baedeker N, Kollaritsch H, Chaplin P. Safety and immunogenicity of modified vaccinia Ankara as a smallpox vaccine in people with atopic dermatitis. Vaccine. 2014 Sep 29;32(43):5696-702. doi: 10.1016/j.vaccine.2014.08.022. Epub 2014 Aug 20. PMID 25149431
- [Result] Darsow U, Sbornik M, Rombold S, Katzer K, von Sonnenburg F, Behrendt H, Ring J. Long-term safety of replication-defective smallpox vaccine (MVA-BN) in atopic eczema and allergic rhinitis. J Eur Acad Dermatol Venereol. 2016 Nov;30(11):1971-1977. doi: 10.1111/jdv.13797. Epub 2016 Jun 29. PMID 27357167